CLINICAL TRIAL: NCT03610243
Title: Use of Patient-centered Self-administered Acupressure for Fatigue Management in Chinese Advanced Cancer Patients: A Randomized Wait-list Controlled Trial
Brief Title: Patient-centered Self-administered Acupressure for Fatigue Management in Chinese Advanced Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW18381
Record Dates: First submitted 2018-07-16; First posted 2018-08-01 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2020-04

CONDITIONS: Advanced Cancer; Acupressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-administered acupressure (Experimental): The proposed self-administered acupressure intervention is patient-centered comprising four pre-selected acupoints that should be applied pressure on by all patients and a list of additional acupoints from which patients can choose two for self-administration according to the personalized recommendations of trainers. In this way, each patient will receive an individualized protocol (four pre-selected and two self-selected acupoints).
  The intervention consists of: individual participant training (Two 2-hour one-on-one training sessions in week 1), self-practice (15 minutes of self-administered acupressure twice a day), and follow-up visits (a 1-hour follow-up visit at weeks 2, 3, and 4).
  Interventions: Behavioral: Self-administered acupressure
- Wait-list control (No Intervention): The wait-list control group will be contacted in the third week to attend a health talk unrelated to symptom management.

INTERVENTIONS:
Behavioral: Self-administered acupressure — Two 2-hour one-on-one training sessions in patient-centered self-administered acupressure will be provided by trainers in the first week (4 hours) in the patient's home or at the university, depending on his/her preference. From the second to fourth weeks of the intervention, participants will engage in 15 minutes of self-administered acupressure twice a day (for a total of 10.5 hours over the 3 weeks). They will log the frequency of self-practice in a diary and be encouraged to undertake self-practice beyond the 4-week intervention. At weeks 2, 3, and 4, a 1-hour follow-up visit will be conducted by the same team of trainers to reinforce learning and self-practice (for a total of 3 hours over the 3 weeks).
  Arms: Self-administered acupressure

SUMMARY:
OBJECTIVE: To evaluate the effect of a patient-centered self-administered acupressure intervention on fatigue, sleep quality, pain, fatigue-sleep disturbance-pain symptom cluster severity, psychological distress, and health-related quality of life among Chinese advanced cancer patients.

HYPOTHESIS TO BE TESTED: Upon intervention completion, the intervention group will exhibit lower levels of fatigue, pain, fatigue-sleep disturbance-pain symptom cluster severity, and psychological distress and higher levels of sleep quality and health-related quality of life than the wait-list control group.

DESIGN and SUBJECTS: A randomized wait-list controlled trial with intervention and wait-list control groups. A total of 30 Chinese advanced cancer patients who screen positive for moderate/severe fatigue with symptoms of insomnia and/or pain will be recruited.

STUDY INSTRUMENTS: Chinese versions of the Brief Fatigue Inventory, Pittsburgh Sleep Quality Index, Brief Pain Inventory, Hospital Anxiety and Depression Scale, Functional Assessment of Cancer Therapy - General, and a demographic questionnaire.

INTERVENTION: A 4-week patient-centered self-administered acupressure intervention comprising 17.5 hours of individual training and self-practice.

MAIN OUTCOME MEASURES: Primary: fatigue. Secondary: sleep quality, pain, fatigue-sleep disturbance-pain symptom cluster severity, psychological distress, health-related quality of life, actigraphy.

DATA ANALYSIS: Linear mixed-effects models to assess between-group differences in outcome measures post-intervention and changes between data collection points, as well as whether the between-group differences vary across time.

EXPECTED RESULTS: The proposed patient-centered self-administered acupressure intervention is useful for alleviating the fatigue and related symptoms experienced by Chinese advanced cancer patients.

DETAILED DESCRIPTION:
The prevalence and impacts of fatigue and related symptoms in cancer patients have been clearly demonstrated in the literature, which also emphasizes the need for evidence-based interventions targeting symptom management in such advanced patients. The main challenge is identifying an intervention that is not only effective in managing cancer-related symptoms but is also feasible, acceptable, and safe for this patient group. The proposed study aims to test the effects of a patient-centered self-administered acupressure intervention on fatigue management for Chinese advanced cancer patients using the robust study design of a randomized, wait-list controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese ethnicity, 18 years of age or older, and ability to communicate in Cantonese or Putonghua;
2. Advanced-stage cancer diagnosis (i.e., colorectum- stage IV; lung - stage IIIB or IV non-small cell or extensive small cell; breast - stage IV; prostate- stage IV; liver - stage IV);
3. An Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1; and
4. Experience of fatigue (rated ≥ 4 on the "fatigue worst" item of the BFI) AND sleep disturbance or pain, or both, in the past week (severity rated ≥ 3 on a 0-10 numeric rating scale)

Exclusion Criteria:

1. are receiving in-patient hospice care; or
2. are taking any medications for insomnia or depression; or
3. have psychiatric or serious medical disorders that may prevent them from comprehending or performing the intervention; or
4. received acupressure or acupuncture in the previous 3 months; or
5. are pregnant or lactating; or
6. have any injury or ulcers around the acupoints

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Brief Fatigue Inventory (BFI) | post-intervention (T1, 4 weeks later)
  The questionnaire will be used for assessing levels of fatigue. The first three items (fatigue severity subscale) ask patients to describe their current fatigue, usual fatigue, and worst fatigue in the past 24 hours, with 0 = "no fatigue" and 10 = "fatigue as bad as you can imagine." The next 6 items (interference subscale) ask the extent to which fatigue interferes with various aspects of life, with 0 = "does not interfere" and 10 = "completely interferes." The mean scores of the 9 items can be categorized as mild (1-3), moderate (4-6), and severe (7-10).
Brief Fatigue Inventory (BFI) | follow-up (T2, 8 weeks after T0)
  The questionnaire will be used for assessing levels of fatigue. The first three items (fatigue severity subscale) ask patients to describe their current fatigue, usual fatigue, and worst fatigue in the past 24 hours, with 0 = "no fatigue" and 10 = "fatigue as bad as you can imagine." The next 6 items (interference subscale) ask the extent to which fatigue interferes with various aspects of life, with 0 = "does not interfere" and 10 = "completely interferes." The mean scores of the 9 items can be categorized as mild (1-3), moderate (4-6), and severe (7-10).

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | pre-intervention (T0, baseline); post-intervention (T1, 4 weeks later); follow-up (T2, 8 weeks after T0)
  This 19-item questionnaire will be used to assess participants' sleep disturbance levels. The items form seven component scores: sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The scores for each component range from 0 to 3 and are summed to produce a global score ranging from 0 to 21, with higher scores denoting poorer sleep quality.
Brief Pain Inventory (BPI) | pre-intervention (T0, baseline); post-intervention (T1, 4 weeks later); follow-up (T2, 8 weeks after T0)
  The pain severity subscale (4 items) will be used to assess participants' pain intensity. The 4-item subscale assesses pain at its "worst," "least," "average," and "now" using an 11-point response format ranging from 0 ("no pain") to 10 ("pain as bad as you can imagine"). Average scores will be calculated and range from 0 to 10. The higher scores refer to higher pain intensity.
Hospital Anxiety and Depression Scale (HADS) | pre-intervention (T0, baseline); post-intervention (T1, 4 weeks later); follow-up (T2, 8 weeks after T0)
  This 14-item questionnaire will be used to measure the severity of participants' psychological distress. Responses are measured on a 4-point scale ranging from 0 ("not present") to 3 ("considerable"). The total score is the sum of the subscale scores (range: 0-42), with a higher score indicating more severe distress.
Functional Assessment of Cancer Therapy - General (FACT-G) | re-intervention (T0, baseline); post-intervention (T1, 4 weeks later); follow-up (T2, 8 weeks after T0)
  The questionnaire consists of 27 items and will be used to assess health-related quality of life. Respondents have to rate each item with a score between 0 ("not at all") and 4 ("very much"). The subscale scores are added to obtain a total score (range=0-108), with a higher score representing a higher level of HRQOL.
Symptom cluster severity | re-intervention (T0, baseline); post-intervention (T1, 4 weeks later); follow-up (T2, 8 weeks after T0)
  the average scores of the BFI and BPI severity subscales and the item on overall sleep quality in the PSQI (to be transformed to a 0-10 scale) will be used. The symptom cluster severity score will be calculated by averaging the fatigue, sleep disturbance, and pain summary scores. The average severity score range from 0 to 10, with higher scores representing higher severity.
Actigraphy | re-intervention (T0, baseline); post-intervention (T1, 4 weeks later); follow-up (T2, 8 weeks after T0)
  Actigraphy will serve as an objective measure of activity levels (fatigue) and sleep quality. Patients will be asked to wear the device for three separate 72-hour periods.

CONTACTS AND LOCATIONS:
Overall Officials: Shuk Ting Cheung, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided